CLINICAL TRIAL: NCT06480851
Title: Effectiveness of Percutaneous Neuromodulation in the Treatment of Cervical Pain in University Students.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Collaborators: Universidad Católica de Ávila (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-026
Record Dates: First submitted 2024-02-03; First posted 2024-06-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain
Keywords: pain; Ecoguided Percutaneous Neuromodulation
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Pain Group (Experimental)
  Interventions: Procedure: Ecoguided Percutaneous Neuromodulation
- Non Neck Pain Group (Active Comparator)
  Interventions: Procedure: Ecoguided Percutaneous Neuromodulation

INTERVENTIONS:
Procedure: Ecoguided Percutaneous Neuromodulation — Ecoguided Percutaneous Neuromodulation over the posterior branch of the cervical multifidus, for 10 minutes, with a frequency of 10 HZ.

SUMMARY:
A non-randomized experimental study will be conducted to investigate the effect of Ecoguided Percutaneous Neuromodulation on patients with and without neck pain in college students. The sample will be collected in a non-probabilistic way at convenience among the students at the San Pablo-CEU University, with a sample that will be divided into two groups: group 1 (G1) with neck pain and group 2 (G2).

ELIGIBILITY:
Inclusion Criteria:

* Current Cervical Pain on a Visual Analog Scale (VAS) greater than 3.
* Neck pain in the last 12 weeks, and no treatment has been performed.
* Disability index of 8% or more on the Neck Disability Index.
* That they have undergone treatment.

Exclusion Criteria:

* Neck pain associated with vertigo.
* Osteoporosis (control X-ray).
* Diagnosed psychological disorders.
* Vertebral fractures (control X-ray).
* Tumors.
* Diagnosed metabolic diseases.
* Neck surgery.
* Belonephobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Pain threshold | up to 1 Week
  Portable hand pressure algometer (FPX 50/220, Wagner Instruments, Greenwich, USA), measured in kg / cm² (kilogram per centimeter squared).

SECONDARY OUTCOMES:
Pain by visual analog scale | Baseline
  usual visual analog scale (VAS) of pain (line from 0: no pain to 10:worst pain)
Pain by visual analog scale | after intervention
  usual visual analog scale (VAS) of pain (line from 0: no pain to 10:worst pain)
Pain by visual analog scale | Follow-up at 1 week
  usual visual analog scale (VAS) of pain (line from 0: no pain to 10:worst pain)
Neck Disability Index Questionnaire. | Baseline
  Quantification of pain and disabilty
Neck Disability Index Questionnaire. | after intervention
  Quantification of pain and disabilty
Neck Disability Index Questionnaire. | Follow-up at 1 week
  Quantification of pain and disabilty
Kinesiophobia | Baseline
  Measured with Tampa Kinesiophobia Scale questionnaire (TSK-11SV) Spanish version. Minimum and maximum values are between 11 and 44 point, a result with higher values indicates higher level of kinesiofobia.
Kinesiophobia | after intervention
  Measured with Tampa Kinesiophobia Scale questionnaire (TSK-11SV) Spanish version. Minimum and maximum values are between 11 and 44 point, a result with higher values indicates higher level of kinesiofobia.
Kinesiophobia | Follow-up at 1 week
  Measured with Tampa Kinesiophobia Scale questionnaire (TSK-11SV) Spanish version. Minimum and maximum values are between 11 and 44 point, a result with higher values indicates higher level of kinesiofobia.
Pain Catastrophizing Scale | Baseline
  Pain Catastrophizing Scale (PAS) will be used to evaluate the participants' pain-related thoughts and feelings.
Pain Catastrophizing Scale | after intervention
  Pain Catastrophizing Scale (PAS) will be used to evaluate the participants' pain-related thoughts and feelings.
Pain Catastrophizing Scale | Follow-up at 1 week
  Pain Catastrophizing Scale (PAS) will be used to evaluate the participants' pain-related thoughts and feelings.
Health-related quality of life | Baseline
  The Short Form Health Questionnaire (SF-36) questionnaire, which examines health-related quality of life under eight sub-titles; It consists of 36 items. The SF36 questionnaire will be used in the study.
Health-related quality of life | after intervention
  The Short Form Health Questionnaire (SF-36) questionnaire, which examines health-related quality of life under eight sub-titles; It consists of 36 items. The SF36 questionnaire will be used in the study.
Health-related quality of life | Follow-up at 1 week
  The Short Form Health Questionnaire (SF-36) questionnaire, which examines health-related quality of life under eight sub-titles; It consists of 36 items. The SF36 questionnaire will be used in the study.
Sonoelastography | Baseline
  This diagnostic test would be executed by a Physiotherapist who has experiences of using General Electric, P9 model ultrasound system for more than three year. The equipment to obtain the image will be used with a frequency of 12 MHz, 22 dB gain, 85 dynamic range, brightness at 17 and depth of 4 cm.
  The transducer will be placed on the spinosa of C4 and the probe will be moved towards the transverse of each of the sides, to identify the image of the multifidus muscle in depth.
  Once the muscle is located in this segment, a longitudinal and transverse image of the muscle will be obtained, performing the elastography at the same time and calculating the elastographic values (tissue resistance in kilopascals and transmission speed in meters/second).
Sonoelastography | after intervention
  This diagnostic test would be executed by a Physiotherapist who has experiences of using General Electric, P9 model ultrasound system for more than three year. The equipment to obtain the image will be used with a frequency of 12 MHz, 22 dB gain, 85 dynamic range, brightness at 17 and depth of 4 cm.
  The transducer will be placed on the spinosa of C4 and the probe will be moved towards the transverse of each of the sides, to identify the image of the multifidus muscle in depth.
  Once the muscle is located in this segment, a longitudinal and transverse image of the muscle will be obtained, performing the elastography at the same time and calculating the elastographic values (tissue resistance in kilopascals and transmission speed in meters/second).
Sonoelastography | Follow-up at 1 week
  This diagnostic test would be executed by a Physiotherapist who has experiences of using General Electric, P9 model ultrasound system for more than three year. The equipment to obtain the image will be used with a frequency of 12 MHz, 22 dB gain, 85 dynamic range, brightness at 17 and depth of 4 cm.
  The transducer will be placed on the spinosa of C4 and the probe will be moved towards the transverse of each of the sides, to identify the image of the multifidus muscle in depth.
  Once the muscle is located in this segment, a longitudinal and transverse image of the muscle will be obtained, performing the elastography at the same time and calculating the elastographic values (tissue resistance in kilopascals and transmission speed in meters/second).

CONTACTS AND LOCATIONS:
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No